CLINICAL TRIAL: NCT06050902
Title: Ultrasound-guided Subclavian Venous Catheterization. A Randomized, Single-blind, Controlled Superiority Trial Comparing Standard Ultrasound Guidance and a New Needle-steering Device
Brief Title: Standard Ultrasound Guidance vs. New Needle-steering Device in Subclavian Venous Catheterization
Acronym: NEEDLEVISIO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NIMAO/2021-1/NB-01
Record Dates: First submitted 2023-09-05; First posted 2023-09-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ultrasound Guidance; Central Venous Catheterization
Keywords: subclavian vein; needle-steering device

STUDY DESIGN:
Intervention Model Description: A randomized, patient- and evaluator-blinded, controlled superiority trial comparing standard ultrasound guidance and a new needle-steering device.
Who Masked: Participant
Masking Description: The patient will be blinded to his or her assignment group. The primary endpoint and secondary endpoints A, D, G, H, will be collected by an assessor independent from the operator, during the central venous catheterization procedure. This assessor will not be blinded to the technique used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard ultrasound guidance for subclavian venipuncture (No Intervention): 62 patients undergoing the usual standard ultrasound guidance technique for subclavian venipuncture
- Subclavian venipuncture using the needle-steering device (Experimental): 62 patients undergoing subclavian venipuncture using the needle-steering device
  Interventions: Device: Subclavian venipuncture for catheter placement using the needle-steering device

INTERVENTIONS:
Device: Subclavian venipuncture for catheter placement using the needle-steering device — 1. Navigation software is implemented in an ultrasound machine.
  2. A linear ultrasound probe (similar in appearance to a standard ultrasound probe) is used
  3. Magnetization of the puncture needle after short introduction of the needle in a dedicated device.
  4. Real time needle guidance on the ultrasound screen during the puncture.
  Arms: Subclavian venipuncture using the needle-steering device

SUMMARY:
Up to two-thirds of intensive care unit patients require central venous catheterization for which ultrasound-guided placement is now recommended. In this context, the team performed a prospective randomized simulation trial on a mannequin ("reduced torso model"), to compare the standard ultrasound guidance technique with an ultrasound-guided technique assisted by a new needle-steering device. The preliminary results show a statistically significant improvement in subclavian venipuncture (shorter success time, fewer multiple skin punctures, fewer punctures of the posterior wall of the subclavian vein and needle redirection, greater comfort) and argue for a clinical trial to test the performance of this new device in situation with intensive care unit patients.

The hypothesis is that the needle-steering device will result in a better success rate of subclavian venous cannulation, at first puncture, compared with the conventional ultrasound-guided technique.

DETAILED DESCRIPTION:
Central venous catheterization is required in up to two-thirds of intensive care unit patients. Ultrasound-guided placement is now recommended over the "blind" technique to decrease the risk of mechanical complications and duration of the procedure. Although the subclavian site is recommended as first-line because of a lower risk of catheter-related infection and thrombosis (than with internal jugular and femoral sites), this approach is underused (< 20% of regular users). There is also a very low use of ultrasound guidance for subclavian catheterization (< 30% of cases), due to technical difficulties such as more complex visualization of the needle.

New magnetic devices theoretically allow better visualization of the needle, a higher success rate and a lower complication rate. In this context, the team performed a prospective randomized simulation trial on a phantom ("reduced torso model"), comparing the standard ultrasound guidance technique with an ultrasound-guided technique assisted by a new needle-steering device in subclavian central venous catheterization (study in progress). The results of this study show a statistically significant improvement in subclavian venipuncture (shorter success time, fewer multiple skin punctures, fewer punctures of the posterior wall of the subclavian vein and needle redirection, greater comfort).

These preliminary results argue for a clinical trial of the practical performance of this new device in intensive care unit patients.

The hypothesis is that the needle-steering device will result in a higher success rate of subclavian venous cannulation at first puncture compared with the conventional ultrasound guidance technique.

ELIGIBILITY:
Inclusion Criteria:

* Any resuscitation patient requiring subclavian venous catheterization.
* Patients or representatives must have given free, informed consent and signed the consent form or patient included in an emergency situation
* Patients must be affiliated to/or beneficiary of a health insurance scheme.
* All patients must be adults (≥18 years of age).

Exclusion Criteria:

* Moribund patients
* Patients with severe primary or secondary hemostasis disorders (Pq < 50 G/L or TP < 30%, or INR > 2).
* Patients with a PaO2/FiO2 ratio < 100 mmHg in mechanically ventilated patients (invasive or non-invasive ventilation).
* Patients with a precarious or unstable respiratory status and significant risk of barotrauma
* Patients for whom it is difficult to visualize the subclavian veins bilaterally (left and right) during ultrasound pre-screening
* Patients with a malformation/deformity of the subclavian region (congenital or acquired: history of surgery/cervical trauma)
* Body mass index < 15 kg/m² ou > 40 kg/m²
* Local infection at the puncture site
* Thrombosis of the subclavian or axillary vein
* Patients participating in a category 1 defined RIPH involving subclavian central venous line placement.
* Patients under court protection, guardianship or curatorship.
* Pregnant, parturient or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-12-26 (Actual); Study Completion 2025-12-26 (Actual)

PRIMARY OUTCOMES:
Successful catheter insertion at first skin puncture: Control group | Day 0
  The main objective is to compare the success rate of subclavian venous cannulation at first puncture between the conventional ultrasound guidance technique and ultrasound guidance assisted by a needle-steering device.
  Successful subclavian venous cannulation (success is defined as catheter insertion at first skin puncture).
  YES/NO
Successful catheter insertion at first skin puncture: Experimental group | Day 0
  The main objective is to compare the success rate of subclavian venous cannulation at first puncture between the conventional ultrasound guidance technique and ultrasound guidance assisted by a needle-steering device.
  Successful subclavian venous cannulation (success is defined as catheter insertion at first skin puncture).
  YES/NO

SECONDARY OUTCOMES:
A. Number of skin punctures required before successful central venous catheterism: Control group | Day 0
  Median number of skin punctures required before successful central venous catheterism. Success is defined as catheter insertion.
A. Number of skin punctures required before successful central venous catheterism: Experimental group | Day 0
  Median number of skin punctures required before successful central venous catheterism. Success is defined as catheter insertion.
B. Complication rate. All causes, composite score: Control group | Day 0
  Onset of at least one complication due to venous puncture. Complications including pneumothorax, arterial puncture, hematoma, malpositioning or puncture failure will all be recorded.
B. Complication rate. All causes, composite score: Control group | Hour 24
  Onset of at least one complication within 24 of venous puncture. Complications including pneumothorax, arterial puncture, hematoma, malpositioning or puncture failure will all be recorded.
B. Complication rate. All causes, composite score: Experimental group | Day 0
  Onset of at least one complication due to venous puncture. Complications including pneumothorax, arterial puncture, hematoma, malpositioning or puncture failure will all be recorded.
B. Complication rate. All causes, composite score: Experimental group | Hour 24
  Onset of at least one complication within 24 of venous puncture. Complications including pneumothorax, arterial puncture, hematoma, malpositioning or puncture failure will all be recorded.
C. Pneumothorax within 24 hours of venous puncture: Control group | Hour 24
  Data collection using a standardized online electronic Case Report Form. Clinical history + frontal chest X-rays taken within one hour of puncture AND at H12-24 +/- ultrasound or computed tomography scan according to clinical or diagnostic doubt (examinations carried out at the discretion of the physicians).
  The number and percentage of patients with pneumothorax will be recorded.
C bis. Drainage required for pneumothorax within 24 hours of venous puncture: Control group | Hour 24
  Data collection using a standardized online electronic Case Report Form. YES/NO
C. Pneumothorax within 24 hours of venous puncture: Experimental group | Hour 24
  Data collection using a standardized online electronic Case Report Form Clinical history + frontal chest X-rays taken within one hour of puncture AND at 12-24 hours +/- ultrasound or computed tomography scan according to clinical or diagnostic doubt (examinations carried out at the discretion of the physicians).
  The number and percentage of patients with pneumothorax will be recorded.
C bis. Drainage required for pneumothorax within 24 hours of venous puncture: Experimental group | Hour 24
  Data collection using a standardized online electronic Case Report Form YES/NO
D. Arterial puncture within 24 hours of venous puncture: Control group | Day 0
  YES / NO Data collection using a standardized online electronic Case Report Form. Any arterial punctures during the procedure will be recorded in numbers and percentages by an independent investigator, present during the procedure and therefore aware of technique used.
D. Arterial puncture within 24 hours of venous puncture: Experimental group | Day 0
  YES / NO Data collection using a standardized online electronic Case Report Form. Any arterial punctures during the procedure will be recorded in numbers and percentages by an independent investigator, present during the procedure and therefore aware of technique used.
E. Hematoma or hemorrhage Grade 3 or over within 24 hours of venous puncture: Control group | Hour 24
  YES / NO. Data collection using a standardized online electronic Case Report Form.
  Clinical history + frontal chest X-rays taken within one hour of puncture AND at H12-24 +/- ultrasound or CT scan according to clinical point of call or diagnostic doubt (examinations carried out according to the choice of the department's physicians).
  Within 24 hours, occurrence of hematoma or hemorrhage grade ≥ 3 (specify whether a therapeutic intervention is required - according to the definition below - or transfusion for intrathoracic bleeding). The occurrence of grade ≥ 3 hematoma or hemorrhage will be established according to the definition of "Common Terminology Criteria for Adverse Events (CTCAE) v5.0": indication for transfusion or invasive intervention (grade 3), need for urgent intervention or alteration of vital prognosis (grade 4), or death (grade 5).
E. Hematoma or hemorrhage Grade 3 or over within 24 hours of venous puncture: Experimental group | Hour 24
  YES / NO. Data collection using a standardized online electronic Case Report Form .
  Clinical history + frontal chest X-rays taken within one hour of puncture AND at H12-24 +/- ultrasound or CT scan according to clinical point of call or diagnostic doubt (examinations carried out according to the choice of the department's physicians).
  Within 24 hours, occurrence of hematoma or hemorrhage grade ≥ 3 (specify whether a therapeutic intervention is required - according to the definition below - or transfusion for intrathoracic bleeding). The occurrence of grade ≥ 3 hematoma or hemorrhage will be established according to the definition of "Common Terminology Criteria for Adverse Events (CTCAE) v5.0": indication for transfusion or invasive intervention (grade 3), need for urgent intervention or alteration of vital prognosis (grade 4), or death (grade 5).
F. Malpositioned catheter seen on the X-ray within 1 hour of venous puncture: Control group | Hour 24
  YES / NO. Data collection using a standardized online electronic Case Report Form .
  Front thoracic radiograph (systematically within one hour of puncture) puncture): "Sweet Spot" technique (approximation of the atriocaval junction, a rectangle in which the position of the lower end of the central venous line: between the lower third of the superior vena cava and the inferior lower edge of the right atrium (located by the cardiophrenic angle). Malpositioning will be recorded as numbers and percentages.
F. Malpositioned catheter seen on the X-ray within 1 hour of venous puncture: Experimental group | Hour 24
  YES / NO. Data collection using a standardized online electronic Case Report Form.
  Front thoracic radiograph (systematically within one hour of puncture) puncture): "Sweet Spot" technique (approximation of the atriocaval junction, a rectangle in which the position of the lower end of the central venous line: between the lower third of the superior vena cava and the inferior lower edge of the right atrium (located by the cardiophrenic angle). Malpositioning will be recorded as numbers and percentages.
G. Time taken from first skin puncture to successful catheter insertion: Control group | Day 0
  In seconds
G. Time taken from first skin puncture to successful catheter insertion: Experimental group | Day 0
  In seconds
H. Failure rate: Control group | Day 0
  Percentage of failures. After three failed punctures, the technique is considered as a failure. Data collection using a standardized online electronic Case Report Form.
  The number of skin punctures will be counted. The criterion "failure" will be retained after 3 unsuccessful skin punctures.
  This requires a change of insertion site and withdrawal from the study. The other complication criteria mentioned above will still be recorded and analyzed but the time will not be collected (criterion G).
H. Failure rate: Experimental group | Day 0
  Percentage of failures. After three failed punctures, the technique is considered as a failure.Percentage of failures. After three failed punctures, the technique is considered as a failure. Data collection using a standardized online electronic Case Report Form.
  The number of skin punctures will be counted. The criterion "failure" will be retained after 3 unsuccessful skin punctures.
  This requires a change of insertion site and withdrawal from the study. The other complication criteria mentioned above will still be recorded and analyzed but the time will not be collected (criterion G).

OTHER OUTCOMES:
Gender | Day 0
  Male/Female
Age | Day 0
  In years
Weight | Day 0
  In kilos
Height | Day 0
  In centimeters
Simplified Severity Index II score | Hour 24
  The SSI II score ( Simplified Severity Index II) is a score used to assess a patient's severity, and is one of the scores used in intensive care and resuscitation. The parameters to be taken into account are the most severe ones collected during the 24 hours following admission to intensive care.
Sequential Organ Failure Assessment score | Day 0
  The Sequential Organ Failure Assessment (SOFA) score is a scoring system that assesses the performance of several organ systems in the body (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) and assigns a score based on the data obtained in each category.
Puncture on right side ? | Day 0
  YES/NO
Patient unconscious ? | Day 0
  YES/NO (absence of contact and movement at the time of puncture)
Positive End Expiratory Pressure | Day 0
  In cm H²O
Indication for central venous catheter : Shock / vasopressor support | Day 0
  YES/NO
Indication for central venous catheter : nutrition | Day 0
  YES/NO
Indication for central venous catheter : Administration of venotoxic drugs | Day 0
  YES/NO
Indication for central venous catheter : Poor venous capital | Day 0
  YES/NO
Indication for central venous catheter : Vascular filling | Day 0
  YES/NO
Indication for central venous catheter : Repeated blood sampling | Day 0
  YES/NO
Indication for central venous catheter : Central venous pressure monitoring | Day 0
  YES/NO

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: Yes
The analysis of the data will be carried out by the BESPIM service of the CHU of Nîmes.
  Within one year after the end of the research or its interruption, a final report will be established and signed by the sponsor and the investigator. This report will be made available to the competent authority. The sponsor will transmit the results of the research in the form of a summary of the final report to the CPP (Comité de Protection des Personnes) and, if necessary, to the ANSM within one year after the end of the research.
Supporting Information: Study Protocol, SAP, ICF, CSR